CLINICAL TRIAL: NCT03402958
Title: General Practitioner's Place in the Treatment of Fracture Osteoporosis in the Elderly
Acronym: GEOFRAGE
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_309_GEOFRAGE
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Osteoporosis is a major public health problem. Its screening and its treatment remain largely insufficient while therapies have demonstrated their effectiveness. In the event of a severe fracture, the update of the 2016/2017 recommendations, prepared by the Research and Information Group on Osteoporosis and the French Rheumatology Society, concerning osteoporosis recommends a specific treatment with bisphosphonates as first-line treatment, without bone densitometry, regardless of age. The frequency of prescribing anti-osteoporotic treatment as an outpatient after a fracture of the upper extremity of the femur is very low (2% to 21% according to the studies). The main factors associated with non-prescription found are co-morbidities (charlson score> 6), dementia, obesity (BMI> 30), chronic alcoholism, male sex, polypharmacy> 4, age. Conversely, the factors associated with prescribing are recurrent falls (> 2 / year), a history of osteoporotic fracture, an Iso Resource Group> 3, female sex, and corticosteroid therapy.

DETAILED DESCRIPTION:
1. / The collection of patients' characteristics upon admission will be based on the computerized patient file and the paper file: socio-demographic data, co-morbidities, functional status, entry / exit treatments, place of residence, source, balance sheet hospital.
2. / Determination with the treating doctor or the pharmacist of the prescriptions of the anti-osteoporotic treatments at 6 months of the hospital care.
3. / Research factors associated with the prescription (or non-prescription) of anti-osteoporotic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 75 or over (hospitalization criteria in the pathway), admitted to the ortho-geriatric ward of the Saint Malo Hospital Center, treated for a fracture of the upper extremity of the femur.

Exclusion Criteria:

* High-energy fracture, pathological fractures (infection, tumor), persons of legal age subject to legal protection (safeguard of justice, guardianship, guardianship), persons deprived of their liberty.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients treated for a fracture of the upper extremity of the femur, included consecutively and retrospectively, during the period of October 2016 - June 2017 at the Saint-Malo Hospital Center
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Frequency of prescription of anti-osteoporosis treatments. | 6 months after surgical management for fracture of the upper end of the femur

SECONDARY OUTCOMES:
Factors associated with the sub-prescription. | Through study completion, an average of 4 months
  The main factors associated with non-prescription found are co-morbidities (charlson score> 6), dementia, obesity (BMI> 30), chronic alcoholism, male sex, polypharmacy> 4, age. Conversely, the factors associated with prescribing are recurrent falls (> 2 / year), a history of osteoporotic fracture, an Iso Resource Group> 3, female sex, and corticosteroid therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Belhomme, Principal Investigator — Rennes University Hospital
Locations (1):
- Hospital Center of Saint-Malo, St-Malo, Britain, France